CLINICAL TRIAL: NCT07397156
Title: 4-Year Mortality, Functional Outcomes, and Quality of Life After ICU-Treated COVID-19-Related ARDS: A Retrospective-Prospective Cohort Study
Brief Title: Long-Term Outcomes After ICU-Treated COVID-19 ARDS
Status: Completed | Type: Observational
Sponsor: University in Zielona Góra (Other)
Responsible Party: Principal Investigator, Jacek Zawadzki, MD PhD, University in Zielona Góra
Other Study IDs: KB 03/165/2021
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: COVID-19; ARDS (Acute Respiratory Distress Syndrome)
Keywords: intensive care unit; ICU survivors; long-term outcomes; 4-year follow-up; health-related quality of life; EQ-5D-5L; modified Medical Research Council (mMRC); Post-COVID-19 Functional Status (PCFS); rehabilitation; return to work; financial burden
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU-Treated COVID-19 ARDS Cohort: Consecutive adult patients treated in the intensive care unit (ICU) for COVID-19-related acute respiratory distress syndrome (ARDS) at a single center in Poland, admitted between December 2020 and July 2021. This was an observational study with no assigned experimental intervention. Long-term vital status was assessed up to approximately 4 years after ICU admission; survivors were invited to a structured telephone follow-up to assess patient-reported outcomes.

SUMMARY:
This observational cohort study describes long-term survival and patient-reported health after intensive care unit (ICU) treatment for COVID-19-related acute respiratory distress syndrome (ARDS) in adults treated in a single center in Poland. The main questions it aims to answer are:

1. What is all-cause mortality up to 4 years after ICU admission for COVID-19-related ARDS?
2. Among long-term survivors, what are the health-related quality of life and functional outcomes approximately 4 years after ICU admission?
3. What rehabilitation use, return-to-work outcomes, and self-reported financial burden are reported during follow-up, and which acute-phase clinical and laboratory factors are associated with late mortality and long-term outcomes?

Participants did not receive any experimental intervention as part of this study. The study team collected clinical information from hospital and ICU records and conducted a structured telephone follow-up with survivors using standardized questionnaires (including EQ-5D-5L for quality of life, the modified Medical Research Council [mMRC] scale for breathlessness, and the Post-COVID-19 Functional Status [PCFS] scale for functional status), as well as questions about rehabilitation and work status.

DETAILED DESCRIPTION:
This is an observational retrospective-prospective cohort study of adults treated in the intensive care unit (ICU) for COVID-19-related acute respiratory distress syndrome (ARDS) at a single center in Poland (University Hospital in Zielona Góra / Temporary COVID-19 Hospital in Zielona Góra). The cohort includes consecutive eligible ICU admissions between December 2020 and July 2021. No experimental intervention was assigned as part of this study.

Acute-phase clinical data were obtained from routinely collected hospital and ICU documentation. These data include baseline demographics, pre-existing comorbidities, severity of illness, and organ dysfunction at ICU admission, selected laboratory and physiological parameters, and key aspects of ICU management and clinical course. Long-term vital status was assessed for approximately 4 years after ICU admission, using available clinical records and follow-up procedures described in the protocol.

A structured telephone follow-up was conducted approximately 4 years after ICU admission among long-term survivors to collect patient-reported outcomes using standardized instruments and a predefined interview script. The follow-up assessment captured health-related quality of life, breathlessness, and functional status, and also included questions on post-discharge rehabilitation, return-to-work status, and self-reported financial burden related to recovery.

Analyses are descriptive and exploratory. Mortality over time is described using time-to-event methods, and associations between selected acute-phase variables and late mortality and long-term patient-reported outcomes are evaluated using multivariable models, with appropriate handling of missing data and sensitivity analyses as specified in the statistical analysis plan. The study was conducted with approval from the relevant ethics committee, and participant consent procedures for the follow-up interview were implemented in accordance with local requirements.

Time perspective: Retrospective extraction of acute-phase ICU data (December 2020-July 2021) with a single structured telephone follow-up of survivors approximately 4 years after ICU admission.

ELIGIBILITY:
Inclusion Criteria:

Baseline cohort (retrospective ICU cohort)

* Adults (≥18 years) admitted to the Temporary Hospital in Zielona Góra ICU between December 2020 and July 2021
* Confirmed SARS-CoV-2 infection
* COVID-19-related acute respiratory distress syndrome (ARDS)
* Required invasive mechanical ventilation during ICU treatment

Prospective follow-up component (telephone interview):

* Confirmed alive at approximately 4 years after ICU admission
* Agreed to participate in a structured telephone interview (voluntary participation)

Exclusion Criteria:

Baseline cohort:

* None (no additional clinical exclusion criteria)

Prospective follow-up component (telephone interview):

* Declined participation in the telephone interview
* Unable to be reached after repeated contact attempts (non-responder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) treated in a single intensive care unit in Poland for COVID-19-related acute respiratory distress syndrome (ARDS) requiring invasive mechanical ventilation during the pandemic surge (December 2020-July 2021). Long-term survival was assessed for the full cohort up to approximately 4 years after ICU admission, and survivors were invited to a structured telephone follow-up to assess patient-reported outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality at 30 Days | 30 days after ICU admission
  Proportion of participants who died from any cause within 30 days of ICU admission.
All-Cause Mortality up to 4 Years | From ICU admission up to 4 years after ICU admission
  Proportion of participants who died from any cause from ICU admission through 4 years after ICU admission (cumulative mortality).

SECONDARY OUTCOMES:
Late All-Cause Mortality Among 30-Day Survivors | Day 31 through 4 years after ICU admission
  Proportion of participants who died from any cause between day 31 and 4 years after ICU admission, among participants alive at day 30.
Health-Related Quality of Life (EQ-5D-5L Index Value) | Approximately 4 years after ICU admission (single telephone follow-up assessment)
  EQ-5D-5L health utility index value derived from the EQ-5D-5L questionnaire administered during structured telephone follow-up.
Self-Rated Health (EQ Visual Analogue Scale [EQ-VAS]) | Approximately 4 years after ICU admission (single telephone follow-up assessment)
  Q-VAS score collected as part of the EQ-5D-5L questionnaire during structured telephone follow-up (among survivors who completed follow-up).
Functional Status (Post-COVID-19 Functional Status [PCFS] Grade) | Approximately 4 years after ICU admission (single telephone follow-up assessment)
  Functional status assessed using the PCFS scale (grade), collected during structured telephone follow-up.
Breathlessness Severity (modified Medical Research Council [mMRC] Score) | Approximately 4 years after ICU admission (single telephone follow-up assessment)
  Breathlessness assessed using the modified Medical Research Council (mMRC) dyspnea scale; reported as mMRC score collected during structured telephone follow-up (among survivors who completed follow-up).
Subjective Cognitive Complaints (Two Screening Items Adapted From the Cognitive Failures Questionnaire [CFQ]) | Approximately 4 years after ICU admission (single telephone follow-up assessment)
  Presence and/or severity of subjective cognitive complaints assessed using two screening items adapted from the Cognitive Failures Questionnaire (CFQ) during structured telephone follow-up (among survivors who completed follow-up).
Sleep Disturbance (Single Screening Item) | Approximately 4 years after ICU admission (single telephone follow-up assessment)
  Self-reported sleep disturbance assessed using a brief single screening item during structured telephone follow-up (among survivors who completed follow-up).
Time to Return to Work | Assessed at approximately 4 years after ICU admission (recall of post-discharge period)
  Self-reported time to return to work after the index hospitalization, collected during structured telephone follow-up (among survivors who were working prior to critical illness and completed follow-up).
Post-Discharge Rehabilitation Exposure and Duration | Assessed at approximately 4 years after ICU admission (recall of post-discharge period)
  Self-reported participation in rehabilitation after hospital discharge and total rehabilitation duration (e.g., weeks), collected during structured telephone follow-up (among survivors who completed follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- University in Zielona Góra, Zielona Góra, Lubusz Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) has not been finalized. Any future sharing would require additional ethics and data protection review and would be considered only in a de-identified form under a data use agreement. Aggregated results will be reported in publications.